CLINICAL TRIAL: NCT00658099
Title: Change in Weight on Insulin Detemir (Levemir®) or Isophane (NPH) Insulin (Insulatard®) in Patients With Type 2 Diabetes Mellitus
Brief Title: Observational Study of Type 2 Diabetes Patients Failing on Oral Anti-diabetic Agents Initiated on Levemir® or Insulatard®
Acronym: EVIDENCE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1976
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: insulin detemir
- B
  Interventions: Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency prescribed by the physician as a result of a normal clinical evaluation
  Groups: A
Drug: insulin NPH — Start dose and frequency prescribed by the physician as a result of a normal clinical evaluation
  Groups: B

SUMMARY:
This trial is conducted in Europe. The aim of this observational study is to evaluate the change in weight in type 2 diabetes patients using Levemir® or Insulatard® under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c greater than 7.0% and/or hypoglycaemia
* variable FBG and/or weight increase
* the selection of the subjects will be at the discretion of the participating physician

Exclusion Criteria:

* non-type 2 diabetes
* current treatment with Levemir® or Insulatard®
* hypersensitivity to Levemir® or Insulatard® or to any of the excipients
* women who are pregnant, breast feeding or have the intention of becoming pregnant within next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes patiens failing on oral anti-diabetic agents
Sampling Method: Non-Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in weight | after 6 months of treatment

SECONDARY OUTCOMES:
The effect on metabolic control assessed by the changes in glycaemic parameters: HbA1c and blood glucose values | after 6 months of treatment
The incidence of hypoglycaemic events | after 6 months of treatment
Safety parameters by collecting (serious) adverse drug reactions, pregnancies and technical complaints. | after 6 months of treatment
The general well-being by using the WHO-5 well-being questionnaire. | after 6 months of treatment
The treatment satisfaction of subjects treated with insulin detemir or NPH insulin by using insulin treatment satisfaction questionnaire | after 6 months of treatment
The satisfaction of physicians who treat the subjects with either insulin detemir or NPH insulin by using 4 questions, which are included in CRF, at the final visit. | after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bucharest, Romania

REFERENCES:
- [Result] Doina Catrinoiu; Effect of Once-Daily Detemir vs NPH Insulin on Body Weight and Metabolic Control When Added to OADs in Type 2 Diabetes; 2029-PO; 69th Scientific Sessions (2009); American Diabetes Association
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com